CLINICAL TRIAL: NCT03502655
Title: Impact of Communication on Pain During Intravenous Cannulation in an Emergency Department: a Randomized Controlled Trial
Brief Title: Discomfort During Intravenous Cannulation in an Emergency Department: Impact of Communication
Acronym: DOUCIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier Hugli (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Olivier Hugli, Head of the inpatient service, Emergency Department, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VVP01112017
Record Dates: First submitted 2017-11-27; First posted 2018-04-19 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Pain, Acute; Catheterization, Peripheral
Keywords: Pain; Peripheral intravenous catheter; Peripheral catheterization; Communication; Emergency Department
MeSH Terms: conditions — Acute Pain; Pain; Communication; Emergencies | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Each eligible patient will be randomized in a 1: 1 ratio between the two arms of the study, double-blind (patient, caregiver, investigator) in the first study and single-blind (patient) in the second study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient allocation to each arm will be based on the sequential opening of an opaque envelope containing an non-consecutive number indicating a track number of the recorded message (control or intervention). Randomization will be based on randomly mixed block of size 2 to 6 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention message (first phase) (Other): Standardized message The intervention will consist in the delivery of a message with a positive content regarding the insertion of the peripheral venous catheter. The message will be delivered through an audio record
  Interventions: Other: Experimental: Intervention message (first phase)
- Control message (first phase) (Active Comparator): Standardized message The intervention will consist in the delivery of a control message, whose content is based upon the usual caregiver-patient communication prior to the insertion of a peripheral venous catheter. The message will be delivered through an audio record.
  Interventions: Other: Placebo Comparator: Control message (first phase)
- Intervention message (second phase) (Other): Standardized message The intervention will consist in the delivery of message with a positive content regarding the insertion of the peripheral venous catheter. The message will be delivered by the health providers themselves before inserting the catheter.
  Interventions: Other: Experimental: Intervention message (second phase)
- Control message (second phase) (Active Comparator): Standardized message In this arm, the patient will be delivered a control message, which content is based upon the usual caregiver-patient communication prior to the insertion of a peripheral venous catheter. The message will be delivered by the caregivers themselves before inserting the catheter.
  Interventions: Other: Placebo Comparator: Control message (second phase)

INTERVENTIONS:
Other: Experimental: Intervention message (first phase) — Effect of positive communication on pain during intravenous cannulation in an emergency department delivered by a recorded message
  Arms: Intervention message (first phase)
Other: Placebo Comparator: Control message (first phase) — Effect of usual communication on pain during intravenous cannulation in an emergency department delivered by a recorded message
  Arms: Control message (first phase)
Other: Experimental: Intervention message (second phase) — Effect of positive communication on pain during intravenous cannulation in an emergency department delivered by a care provider
  Arms: Intervention message (second phase)
Other: Placebo Comparator: Control message (second phase) — Effect of usual communication on pain during intravenous cannulation in an emergency department delivered by a care provider
  Arms: Control message (second phase)

SUMMARY:
The main goal of this study is to investigate whether the communication between patients and healthcare providers has an impact on pain and anxiety induced by the insertion of a peripheral venous catheter in an emergency department. Another goal is to determine if the effect is mediated by the content of the message in itself or if it is mediated by non-verbal cues . Therefore, the message will be delivered by either an audio recording in the first phase of the study, and by the healthcare providers themselves in the second phase of the study. A secondary goal is to assess whether there are discrepancies between the patients' pain and anxiety reports and the healthcare providers' evaluation of the patient's pain and anxiety.

DETAILED DESCRIPTION:
A medical or surgical emergency is a stressful life event. An emergency department is also a noisy and sometimes chaotic environment, contributing in itself to increase the anxiety related to the primary cause of the emergency consultation. Some common medical procedures, such as placing an intravenous catheter, may not only induce pain, but may exacerbate patients' anxiety or pre-existing pain. The well-being of patients, especially during invasive medical procedures, can however be improved by various communication techniques. However, the medical literature and clinical observation have shown that negative words are traditionally used to warn patients of an impending painful stimulus. However, contrary to common beliefs and practices, this type of warning can increase pain and anxiety. Using words with negative emotional content has an even greater impact than the positive impact of using words with positive emotional content. However, studies that have explored the impact of such messages suffer from two limitations: first, they were not conducted in the context of emergency department, and second, the effect attributable to healthcare providers themselves was not studied. However, healthcare providers who deliver a message with a positive or negative content in the context of a study are not blinded to message, therefore are aware of the arm of the intervention. This lack of double-blinding may introduces a bias, namely that the benefit of a positive message can be linked to healthcare providers and their global interaction with patients, and not just to verbal content. of the message. It is indeed possible that the caregivers, in a more or less conscious way, add in their communication elements congruent with the message studied, whether in the field of verbal or nonverbal communication (tone of voice, warmth, empathy , etc.).

The purpose of this study is therefore to investigate whether the modulation of information relating to the setting up of a CIP in emergencies has an impact on patients' pain and their level of anxiety. It also seeks to determine if this effect is comparable, whether the message is delivered by a standardized audio recording or by caregivers. Finally, it aims to explore whether there are differences in the assessment of pain and anxiety made by patients and that made by caregivers.

Statistical analysis will be realized using the Stata software, version 14 (StataCorp, Tx, USA). Descriptive data will be presented by mean and standard deviation, median and interquartile space or proportions regarding continuous gaussian, non-gaussian and categorical variables. Comparison between randomized groups will be done by using non paired Student t-test or Wilcoxon rank sum test regarding continuous variables, and by Chi2 test or Fisher exact regarding categorical variables, according to what is appropriate.

This study aims to demonstrate the superiority of an informative message with positive content over pain perception during intravenous cannulation. Statistical power is set at 80% to prove a difference, with alpha threshold at 0.05. Mean pain intensity is estimated at 34 mm on a Visual Analog Scale (possible intensity from 0 to 100 mm), with an estimated standard deviation at 24 mm. To detect the smallest clinically significative decrease in pain intensity (13 mm) caused by the intervention, a sample of 110 patients, that is 55 patients per group, is needed. Taking missing data or post-randomization patient withdrawal (estimated at 10%) into account, 60 patients will be randomized per group. A minimum of 240 patients in total for the two phases (that is the four arms of the study) will be needed to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or more;
* Patient whose medical care requires a peripheral venous catheter;
* Insertion of the peripheral venous catheter on the upper limb.

Exclusion Criteria:

* Patient clinically unstable;
* Patient incapable of discernment or with whom it is difficult to communicate (altered mental status, intoxication, alcoholized patient, insufficient French notions to give an informed consent and answer questions about pain and anxiety, hearing-impaired patient);
* Patient unable to correctly use the rulers (e.g. visually impaired patient);
* Impaired upper limb (e.g. lymphedema);
* Patient incarcerated;
* Patient transferred from another hospital;
* Patient who has already taken part in the study;
* Patient who knows beforehand that communication will be evaluated;
* Patient, caregiver or investigator who knows beforehand which message will be delivered (first phase of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Patients' self-evaluation of pain intensity and pain unpleasantness before the peripheral venous catheter's insertion (basal rates). | Pain intensity and unpleasantness will be assessed immediately at the end of the procedure.
  Pain intensity and unpleasantness will be assessed via specifically created Visual Analog Scales on a small ruler. This ruler will be presented to the patients who will place the slider on a line going from one extreme to the other (no pain / worst pain imaginable) and corresponding, on their other side, to a value between 0 and 100 mm on a 100 mm long line. This numerical value measured in millimeters will be reported in the CRF by the co-investigators.
Patients' self-evaluation of pain intensity and pain unpleasantness due to the insertion of a peripheral venous catheter. | Pain intensity and unpleasantness due to the catheter's insertion will be assessed about two minutes after the peripheral venous catheter's insertion.
  Pain intensity and unpleasantness will be assessed via specifically created Visual Analog Scales on a small ruler. This ruler will be presented to the patients who will place the slider on a line going from one extreme to the other (no pain / worst pain imaginable) and corresponding, on their other side, to a value between 0 and 100 mm on a 100 mm long line. This numerical value measured in millimeters will be reported in the CRF by the co-investigators.

SECONDARY OUTCOMES:
Patients' self-evaluation of anxiety before the peripheral venous catheter's insertion (basal rate). | Anxiety will be assessed about ten minutes before the peripheral venous catheter's insertion.
  Anxiety will be assessed via specifically created Visual Analog Scales on a small ruler. This ruler will be presented to the patients who will place the slider on a line going from one extreme to the other (no anxiety at all / extremely anxious) and corresponding, on their other side, to a value between 0 and 100 mm on a 100 mm long line. This numerical value measured in millimeters will be reported in the CRF by the co-investigators.
Patients' self-evaluation of anxiety after the peripheral venous catheter's insertion. | Anxiety will be assessed about two minutes after the peripheral venous catheter's insertion.
  Anxiety will be assessed via specifically created Visual Analog Scales on a small ruler. This ruler will be presented to the patients who will place the slider on a line going from one extreme to the other (no anxiety at all / extremely anxious) and corresponding, on their other side, to a value between 0 and 100 mm on a 100 mm long line. This numerical value measured in millimeters will be reported in the CRF by the co-investigators.
Caregivers' evaluation of patients' pain intensity, pain unpleasantness and anxiety. | Caregivers' evaluation of patients' pain intensity, pain unpleasantness and anxiety will be assessed about ten minutes after the insertion of the peripheral venous catheter.
  Patients' pain intensity, pain unpleasantness and anxiety, as evaluated by the caregivers, will be assessed using specifically created Visual Analogue Scales, similar to the patients' scales only in paper form. The caregivers will indicate their evaluation by tracing a line on the scale going from one extreme to the other (no pain / worst pain imaginable). The co-investigators will then measure the distance between no pain (i.e. 0) and the line traced by the caregiver in millimeters and report this numerical value in the CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hugli, PD-MER, MPH, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaptchuk TJ, Kelley JM, Conboy LA, Davis RB, Kerr CE, Jacobson EE, Kirsch I, Schyner RN, Nam BH, Nguyen LT, Park M, Rivers AL, McManus C, Kokkotou E, Drossman DA, Goldman P, Lembo AJ. Components of placebo effect: randomised controlled trial in patients with irritable bowel syndrome. BMJ. 2008 May 3;336(7651):999-1003. doi: 10.1136/bmj.39524.439618.25. Epub 2008 Apr 3. PMID 18390493
- [Background] Krauss BS. "This may hurt": predictions in procedural disclosure may do harm. BMJ. 2015 Feb 6;350:h649. doi: 10.1136/bmj.h649. PMID 25663166
- [Background] Lang EV, Tan G, Amihai I, Jensen MP. Analyzing acute procedural pain in clinical trials. Pain. 2014 Jul;155(7):1365-1373. doi: 10.1016/j.pain.2014.04.013. Epub 2014 Apr 13. PMID 24731852
- [Background] Li SF, Greenwald PW, Gennis P, Bijur PE, Gallagher EJ. Effect of age on acute pain perception of a standardized stimulus in the emergency department. Ann Emerg Med. 2001 Dec;38(6):644-7. doi: 10.1067/mem.2001.119849. PMID 11719743
- [Background] Nevin K. Influence of sex on pain assessment and management. Ann Emerg Med. 1996 Apr;27(4):424-6. doi: 10.1016/s0196-0644(96)70222-6. No abstract available. PMID 8604851
- [Background] Page MG, Katz J, Stinson J, Isaac L, Martin-Pichora AL, Campbell F. Validation of the numerical rating scale for pain intensity and unpleasantness in pediatric acute postoperative pain: sensitivity to change over time. J Pain. 2012 Apr;13(4):359-69. doi: 10.1016/j.jpain.2011.12.010. Epub 2012 Mar 15. PMID 22424915
- [Background] Rat P, Jouve E, Pickering G, Donnarel L, Nguyen L, Michel M, Capriz-Ribiere F, Lefebvre-Chapiro S, Gauquelin F, Bonin-Guillaume S. Validation of an acute pain-behavior scale for older persons with inability to communicate verbally: Algoplus. Eur J Pain. 2011 Feb;15(2):198.e1-198.e10. doi: 10.1016/j.ejpain.2010.06.012. Epub 2010 Jul 17. PMID 20638878
- [Background] Singer AJ, Richman PB, Kowalska A, Thode HC Jr. Comparison of patient and practitioner assessments of pain from commonly performed emergency department procedures. Ann Emerg Med. 1999 Jun;33(6):652-8. PMID 10339680
- [Background] Wells RE, Kaptchuk TJ. To tell the truth, the whole truth, may do patients harm: the problem of the nocebo effect for informed consent. Am J Bioeth. 2012;12(3):22-9. doi: 10.1080/15265161.2011.652798. PMID 22416745
- [Result] Dutt-Gupta J, Bown T, Cyna AM. Effect of communication on pain during intravenous cannulation: a randomized controlled trial. Br J Anaesth. 2007 Dec;99(6):871-5. doi: 10.1093/bja/aem308. Epub 2007 Oct 30. PMID 17977860
- [Result] Greville-Harris M, Dieppe P. Bad is more powerful than good: the nocebo response in medical consultations. Am J Med. 2015 Feb;128(2):126-9. doi: 10.1016/j.amjmed.2014.08.031. Epub 2014 Sep 16. PMID 25232716
- [Result] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Result] Lang EV, Hatsiopoulou O, Koch T, Berbaum K, Lutgendorf S, Kettenmann E, Logan H, Kaptchuk TJ. Can words hurt? Patient-provider interactions during invasive procedures. Pain. 2005 Mar;114(1-2):303-9. doi: 10.1016/j.pain.2004.12.028. Epub 2005 Jan 26. PMID 15733657
- [Result] Mistiaen P, van Osch M, van Vliet L, Howick J, Bishop FL, Di Blasi Z, Bensing J, van Dulmen S. The effect of patient-practitioner communication on pain: a systematic review. Eur J Pain. 2016 May;20(5):675-88. doi: 10.1002/ejp.797. Epub 2015 Oct 22. PMID 26492629
- [Result] Varelmann D, Pancaro C, Cappiello EC, Camann WR. Nocebo-induced hyperalgesia during local anesthetic injection. Anesth Analg. 2010 Mar 1;110(3):868-70. doi: 10.1213/ANE.0b013e3181cc5727. Epub 2009 Dec 30. PMID 20042440
- [Result] Wang F, Shen X, Xu S, Liu Y, Ma L, Zhao Q, Fu D, Pan Q, Feng S, Li X. Negative words on surgical wards result in therapeutic failure of patient-controlled analgesia and further release of cortisol after abdominal surgeries. Minerva Anestesiol. 2008 Jul-Aug;74(7-8):353-65. PMID 18612266
- [Derived] Berna C, Favre-Bulle A, Bonzon A, Gross N, Gonthier A, Gerhard-Donnet H, Taffe P, Hugli O. Is Positive Communication Sufficient to Modulate Procedural Pain and Anxiety in the Emergency Department? A Randomized Controlled Trial. Psychosom Med. 2023 Nov-Dec 01;85(9):772-777. doi: 10.1097/PSY.0000000000001246. Epub 2023 Aug 24. PMID 37678374

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT03502655/Prot_SAP_000.pdf